CLINICAL TRIAL: NCT03540264
Title: Tooth Wear : Diagnosis- Treatment Decision- Management- Monitoring- Randomized Clinical Trial
Brief Title: Tooth Wear:m Tooth Wear : Diagnosis- Treatment Decision
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017/24NOV/531
Record Dates: First submitted 2018-03-05; First posted 2018-05-30 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Dental Wear
MeSH Terms: conditions — Tooth Wear

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The statistician will be blind to the treatment assigned to indivivual patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Composite resin (Active Comparator): Restoration with composite resin has shown good clinical performance and limited occlusal wear. The Clearfil Majesty will be used in the present study.
  Interventions: Device: Clearfil Majesty TM
- Polymer-infiltrated-ceramic-network (Active Comparator): This hybrid material seems to be a promising material that imitates natural tooth properties. The VITA-Enamic® will be used in this study.
  Interventions: Device: Vita-Enamic®

INTERVENTIONS:
Device: Clearfil Majesty TM — Tooth wear - composite resin
  Arms: Composite resin
Device: Vita-Enamic® — Tooth wear - polymer-infiltrated-ceramic-network
  Arms: Polymer-infiltrated-ceramic-network

SUMMARY:
Tooth wear is a physiological process occurring from normal functioning of the dentition throughout lifetime.

DETAILED DESCRIPTION:
The studies in the current literature indicated that both techniques of tooth preparation and the materials used are appropriate for the treatment of this condition, but the tendency is to reduce tooth preparation as reasonably possible. In this clinical trial, the investigators will compare the outcomes of direct resin composite and indirect polymer-infiltrated-ceramic-network.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older, in good general health, willing to participate in the study and accepting to come to regular controls in the future.
* Patients representing any type of significant tooth wear (≥ 1 mm depth) with dentine exposure in at least 4 teeth: localized tooth wear anterior or posterior teeth and generalized tooth wear anterio and posterior teeth.
* Patients having posterior support with at least 4 molars in occlusion, 1 pair per side, excluding third molar.

Exclusion Criteria:

* Patients wearing removable partial prosthesis
* Patients presenting skeletal Cl III occlusal Relationship
* Patients with remaining clinical crown of ≤ 3 mm in height and presenting tooth anomaly in shape and number in addition to anterior diastemas.
* Patients with symptomatic temporomandibular joint disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2018-02-26 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Restoration | up to 3 years
  by modified USPHS criteria

CONTACTS AND LOCATIONS:
Overall Officials: De Carvalho Joana, Dentist, Pr, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium